CLINICAL TRIAL: NCT03297151
Title: The Effect of Milk Derived Protein Supplementation on Muscle Recovery Following Resistance Exercise
Brief Title: Protein Supplementation and Recovery of Muscle Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: FHIHAPN3.3RX; TC20130001 (Other Grant/Funding Number: Enterprise Ireland)
Record Dates: First submitted 2017-08-17; First posted 2017-09-29 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Resistance Training; Muscle Damage
Keywords: Resistance Training; Muscle Function; Protein Synthesis
MeSH Terms: interventions — Whey

STUDY DESIGN:
Intervention Model Description: Block randomised, between group study
Who Masked: Participant, Investigator
Masking Description: Double blind (participant and investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL (Sham Comparator): Intervention: Dietary Supplement: Non-essential amino acids A group of subjects ingesting a liquid beverage (per kilogram body mass: 0.33g non-essential amino acids dissolved in water ) prior to completion of a prescribed resistance exercise training (RET) session.
  Muscle Contractile Function to be conducted prior to and following the RET session by laboratory-based ergometry.
  Muscle Protein Synthesis induced by RET to be measured by deuterium incorporation in to skeletal muscle sampled by microbiopsy.
  Interventions: Dietary Supplement: CONTROL
- PROTEIN (Active Comparator): Intervention: Dietary Supplement: Whey Protein Concentrate A group of subjects ingesting a liquid beverage (per kilogram body mass: 0.33g of Whey Protein Concentrate dissolved in water ) prior to completion of a prescribed resistance exercise training (RET) session.
  Muscle Contractile Function to be conducted prior to and following the RET session by laboratory-based ergometry. Muscle Protein Synthesis induced by RET to be measured by deuterium incorporation in to skeletal muscle sampled by microbiopsy.
  Interventions: Dietary Supplement: Whey Protein Concentrate
- HYDROLYSATE (Active Comparator): Intervention: Dietary Supplement: Whey Protein Hydrolysate A group of subjects ingesting a liquid beverage (per kilogram body mass: 0.33g of Whey Protein Hydrolysate dissolved in water ) prior to completion of a prescribed resistance exercise training (RET) session.
  Muscle Contractile Function to be conducted prior to and following the RET session by laboratory-based ergometry. Muscle Protein Synthesis induced by RET to be measured by deuterium incorporation in to skeletal muscle sampled by microbiopsy.
  Interventions: Dietary Supplement: Whey Protein Hydrolysate

INTERVENTIONS:
Dietary Supplement: CONTROL — Food grade mixture of non-essential amino acids in powdered form, flavoured and instantised to be dissolved in water.
  Supplied by Carbery Food Ingredients Limited, Ballineen, Ireland. Product Reference Number 10955
  Arms: CONTROL
Dietary Supplement: Whey Protein Concentrate — Whey protein concentrate in powdered form, flavoured and instantised to be dissolved in water.
  Supplied by Carbery Food Ingredients Limited, Ballineen, Ireland. Trade name of product is Carbelac80 Instant Product Reference Number 10431
  Other Names: Carbelac80 Instant
  Arms: PROTEIN
Dietary Supplement: Whey Protein Hydrolysate — Whey protein concentrate hydrolysate (degree of hydrolysate 27%) in powdered form, flavoured and instantised to be dissolved in water.
  Supplied by Carbery Food Ingredients Limited, Ballineen, Ireland. Product Reference Number 10468
  Arms: HYDROLYSATE

SUMMARY:
The focus is performance nutrition. Resistance exercise can induce low level muscle damage in conjunction with impaired contractile function. Milk-derived proteins contain, or induce, bioactive properties that assist muscle recovery and restore/improve muscle function. The aim of the research is the recovery of muscle function following resistance exercise.

In this study, the investigators propose to undertake a comparison of the ingestion of two milk-derived protein-based recovery drinks on muscle function after resistance exercise compares to an isonitrogenous, non-essential amino acid control.

DETAILED DESCRIPTION:
Study Design: A block randomised design of 3 groups of resistance-exercise trained (RET) men

Participants: 24 young, healthy, resistance exercise trained, males aged 18 - 35 years.

Recovery drinks; CONTROL - an isonitrogenous, non-essential amino acid solution; PROTEIN - a milk-based whey protein concentrate (WPC), WPC-80; HYDROLYSATE - a hydrolysed derivative of WPC-80.

Day 1, Pre-screening consisting of:

* medical history and examination by a clinician
* blood sample to be evaluated for health-related contraindications
* body composition measurement by dual energy x-ray absorptiometry (DXA) to determine whole body and segmental lean tissue mass;
* exercise training log (6 month recall);
* dietary consultation;
* habitual physical activity level assessed by European Physical Activity Questionaire (EPAQ)-2

Day 2 - 8: Participants will be "free-living" during this time. Participants will record dietary intake under the guidance of a qualified dietitian and sports nutritionist.

Day 9 and 10: Participants will complete two familiarisation sessions to the resistance exercise and muscle function testing procedures.

A single blood sample (5ml) will be drawn following o/n fast on each day. On day 2 participants will drink a metered dose of deuterated water (around 200ml) containing deuterium. A saliva sample will be taken before and after consuming this bolus.

Day 11-17. During this experimental phase diet is prescribed and provided. The diet is based on habitual food intake standardized to body mass.

Day 11: O/n fasted blood, saliva and 1st micro-biopsy of muscle obtained; Muscle function measured prior to and upon completion of a prescribed bout of resistance exercise training (RET); The recovery drink (0.33 g protein/kg body mass) is ingested; 3 hours following completion of RET a 2nd micro-biopsy of muscle is obtained.

Day 12: O/n fasted blood and saliva is obtained Muscle function measured and recovery drink (0.33 g protein/kg body mass) consumed.

Day 13: O/n fasted blood and saliva is obtained Muscle function measured followed by the 2nd RET bout and recovery drink (0.33 g protein/kg body mass) consumed.

Day 14: O/n fasted blood and saliva is obtained Muscle function measured and recovery drink (0.33 g protein/kg body mass) consumed.

Day 15: O/n fasted blood and saliva is obtained Muscle function measured followed by the 3rd RET bout and recovery drink (0.33 g protein/kg body mass) consumed.

Day 16 O/n fasted blood, saliva and 3rd micro-biopsy of muscle obtained Muscle function measured and recovery drink (0.33 g protein/kg body mass) consumed.

Day 17: O/n fasted blood and saliva is obtained Muscle function measured

ELIGIBILITY:
Inclusion Criteria:

* risk
* no known current illness or physically active
* resistance-exercise trained
* no known intolerance to milk-based products
* no known blood born disease or medication that would adversely affect participation
* no adverse risk to venepuncture

Exclusion Criteria:

• recent musculoskeletal injury

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Change in Muscle Contractile Function | Day 9, 10, 11, 12, 13, 14, 15, 16 and 17
  Maximal Voluntary Contract (MVC) of Knee Extensor Muscle measured by laboratory-based ergometry

SECONDARY OUTCOMES:
Change in Muscle Protein Synthesis | Day 11 and 16
  The fractional rate of muscle protein synthesis (MPS) measured by deuterium incorporation into skeletal muscle sampled by microbiopsy

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Jakeman, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Co Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Food For Health Ireland National Technology Centre — http://FHI.ie

DOCUMENTS (2):
  • Study Protocol (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT03297151/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT03297151/SAP_001.pdf